CLINICAL TRIAL: NCT06924918
Title: Scalp Acupuncture Treatment for Chronic Tic Disorders in Children: A Multicenter Randomized Controlled Trial
Brief Title: Scalp Acupuncture Treatment for Chronic Tic Disorders in Children
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Fudan University (Other)
Responsible Party: Principal Investigator, wangjun, Deputy Director of the Department, Children's Hospital of Fudan University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CHFudanU2025-29
Record Dates: First submitted 2025-04-05; First posted 2025-04-13 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Tic Disorder
Keywords: Tic Disorder; scalp acupuncture treatment; Multicenter Randomized Controlled Trial
MeSH Terms: conditions — Tic Disorders

STUDY DESIGN:
Intervention Model Description: This is an outcome assessor and data analyst-blinded, randomized, controlled superiority trial.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Data analyst
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Scalp Acupuncture Treatment Group (Experimental): This group will receive scalp acupuncture treatment combined with Tuina treatment. The scalp acupuncture treatment and Tuina treatment will be implemented two times a week, eight times per treatment course, with each patient having three treatment courses in total.
  Interventions: Other: Scalp Acupuncture Treatment; Other: Tuina Treatment Group
- Tuina Treatment Group (Active Comparator): This group will receive Tuina treatment only. The Tuina treatment will be implemented two times a week, eight times per treatment course, with each patient having three treatment courses in total.
  Interventions: Other: Tuina Treatment Group

INTERVENTIONS:
Other: Scalp Acupuncture Treatment — Acupoint Selection:
  Baihui (GV20), Sishencong (EX-HN1), Frontal Midline Line (MS1), Vertex Midline Line (MS5), Lateral Line 1 of Vertex (MS7), Shenting (GV24), Yintang (EX-HN3), Shuaigu (GB8)
  Acupuncture Manipulation:
  Needles with a diameter of 0.18-0.35 mm and length of 13-25 mm are selected. After routine disinfection of the acupoint skin, the practitioner holds the micro-needle and quickly inserts it into the subcutaneous tissue at an insertion angle of 15°-30°, primarily using superficial horizontal insertion. The insertion depth is maintained at 15-20 mm, adjusted according to the child's head circumference, body size, and body mass. Needles are retained for 30 minutes.
  Course of treatment:
  2 times a week for 12 weeks
  Arms: Scalp Acupuncture Treatment Group
Other: Tuina Treatment Group — Prescription:
  Spleen Meridian (Pi Jing), Small Heavenly Heart (Xiao Tianxin), Five Finger Joints (Wu Zhi Jie), Internal Bagua (Nei Bagua), Hand Yin-Yang (Shou Yin Yang), Upper Three Passes (Shang San Guan), Gushing Spring (Yongquan, KI-1), Leg Three Miles (Zusanli, ST-36) Manipulation Techniques
  Pushing/Kneading the Spleen Meridian (Tonifying Pi Jing):
  Tapping Small Heavenly Heart (Xiao Tianxin):
  Kneading the Five Finger Joints (Wu Zhi Jie):
  Moving the Internal Bagua (Nei Bagua):
  Separating Yin and Yang (Separating Shou Yin Yang):
  Pushing Up the Upper Three Passes (Pushing San Guan):
  Kneading Gushing Spring (Yongquan, KI-1):
  Kneading Leg Three Miles (Zusanli, ST-36):
  2 times a week for 12 weeks

SUMMARY:
The goal of this clinical trial is to learn if scalp acupuncture works to treat chronic tic disorders (CTD) in children. It will also learn about the safety of scalp acupuncture. The main questions it aims to answer are:

* Does scalp acupuncture improve clinical symptoms and social functioning, and enhance quality of life in children with chronic tic disorders?
* Researchers will compare scalp acupuncture combined with Tuina treatment to Tuina treatment to see if scalp acupuncture treatment works to treat scalp acupuncture.

Participants will:

* Receive scalp acupuncture treatment and Tuina treatment for 2 times per week and last for 12 weeks.
* Receive questionnaire survey using the following scales: the Yale Global Tic Severity Scale (YGTSS), the Clinical Global Impression (CGI) Scale, the Children and Adolescents Quality of Life Scale for Tourette Syndrome (C&A-GTS-QOL) and the Child Behavior Checklist (CBCL).

DETAILED DESCRIPTION:
Tourette Disorder (TD), which includes Temporary Tic Disorder (TTD), Chronic Motor or Vocal Tic Disorder (CTD), and Tourette Syndrome (TS), is a common neuropsychiatric condition in children and teenagers. It is characterized by sudden, rapid, repetitive, and non-rhythmic movements (motor tics) or sounds (vocal tics), or both. TD is most common in school-aged children, typically starting between ages 3 and 15, with symptoms peaking around ages 10-12. Children with TD often experience other challenges like obsessive-compulsive behaviors (OCD), attention-deficit hyperactivity disorder (ADHD), autism spectrum traits, anxiety, depression, sleep issues, or self-harm. These challenges can significantly impact the child's life, family, and society, making TD a chronic and difficult-to-treat condition that affects young people's health and quality of life.

Current treatments mainly involve medications and behavioral therapy. Drugs are often the first choice and can help reduce core symptoms, but side effects, poor long-term adherence, and symptom relapse after stopping medication make many families hesitant to use them. Behavioral therapy has fewer side effects but requires long-term effort, works slowly, and may not suit younger children.

Traditional acupuncture has shown promise in treating childhood neuropsychiatric conditions. Research suggests acupuncture may help by regulating nervous system function, improving brain blood flow, and balancing brain chemicals. Recent studies on TD report that acupuncture might reduce tic frequency/severity, improve mood/behavior, and enhance daily life. However, reviews of existing research point out flaws like small study groups, poorly designed methods, and lack of proper control groups. These issues create uncertainty about acupuncture's true effectiveness for TD, highlighting the need for larger, better-designed studies to confirm its benefits.

In this 12-week, randomized, controlled trial with outcome assessor and data analyst blinding, a total of 136 children with chronic tic disorders (CTD) will be enrolled. Participants will be randomly allocated into two groups: 1) the scalp acupuncture group (n = 68), which will receive scalp acupuncture combined with Tuina treatment (two sessions per week for 12 weeks), and 2) the routine intervention control group (n = 68), which will undergo Tuina treatment. Assessments will be conducted at baseline, weeks 4, 8, and 12 (treatment phase), and week 24 (follow-up phase) using the Yale Global Tic Severity Scale (YGTSS), Clinical Global Impression (CGI) scale, Children and Adolescents' Quality of Life Scale for Gilles de la Tourette Syndrome (C&A-GTS-QOL) and Child Behavior Checklist (CBCL).

The study will be conducted across five clinical centers: the Children's Hospital of Fudan University, Xiamen Children's Hospital, First People's Hospital of Zunyi, The Second Affiliated Hospital of Guizhou University of Traditional Chinese Medicine and Dehong Prefecture People's Hospital.

ELIGIBILITY:
Inclusion Criteria:

1. Meet the diagnostic criteria for Chronic Motor Tic Disorder or Vocal Tic Disorder as defined by the DSM-5 (Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition), confirmed by at least one associate chief psychiatrist. Tic severity must be mild to moderate (YGTSS total score ≤50).
2. Age: 4-12 years old.
3. Patients with comorbid conditions (e.g., ADHD, OCD, oppositional defiant disorder, depression, anxiety) must have stable medication regimens with no anticipated adjustments during the study period.
4. Patients currently taking traditional Chinese herbal medications or decoctions for tics must agree to discontinue use and complete a 2-4 week washout period before enrollment.
5. Newly diagnosed cases unwilling to start medication, patients with unsatisfactory medication-controlled tics, or those reporting significant side effects are eligible if tics have remained stable (unchanged for ≥2 months) without improvement.
6. Voluntary participation with a signed informed consent form.

Exclusion Criteria:

1. IQ（intelligence quotient） ≤80.
2. Severe cardiac, liver, kidney diseases, hyperthyroidism, or unstable vital signs.
3. Comorbid conditions such as intellectual disability, autism spectrum disorder, childhood schizophrenia, bipolar disorder, specific learning disorders, or epilepsy.
4. Patients currently taking traditional Chinese herbal medications or decoctions for tics who refuse to discontinue use.
5. Patients unable to tolerate acupuncture therapy.
6. Prior acupuncture treatment for tics proven ineffective.

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 136 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Yale Global Tic Severity Scale (YGTSS) | Assessments will be conducted at baseline, during the treatment phase (weeks 4, 8, and 12), and during the follow-up phase (week 24).
  Yale Global Tic Severity Scale (YGTSS) is a standardized instrument designed to assess the severity of tic disorders. It evaluates motor tics and vocal tics separately across five dimensions: frequency, intensity, complexity, interference, and overall severity, with each dimension scored on a scale of 0-5 points. The total scores for motor and vocal tics range from 0-25 points each. Additionally, the YGTSS assesses the overall functional impairment caused by tics in daily life, social interactions, academic performance, and occupational activities, with impairment scores ranging from 0-50 points. Total YGTSS Score is calculated as the sum of motor tic score, vocal tic score, and functional impairment score, yielding a composite score of 0-100 points, where higher scores indicate greater symptom severity.

SECONDARY OUTCOMES:
Clinical Global Impression (CGI) Scale | Assessments will be conducted at baseline, during the treatment phase (weeks 4, 8, and 12), and during the follow-up phase (week 24).
  Clinical Global Impression (CGI) Scale, a globally recognized efficacy assessment tool for psychiatric disorders, comprises three domains: Severity of Illness (CGI-S), Global Improvement (CGI-I), and Efficacy Index (CGI-E). For this study, only CGI-S and CGI-I will be utilized.
  CGI-S evaluates the relative severity of current psychiatric symptoms based on clinical expertise, rated on a 7-point scale:
  1: No illness 7: Extremely severe illness Higher scores indicate greater symptom severity.
  CGI-I assesses overall clinical improvement following intervention, scored on a 7-point scale ranging from -2 (very marked worsening) to +4 (very marked improvement), with 0 indicating no change.By integrating CGI-S (baseline severity) and CGI-I (post-treatment change), this scale provides a structured framework to objectively quantify disease burden and therapeutic response in patients with tic disorders following acupuncture intervention.
Children and Adolescents Quality of Life Scale for Tourette Syndrome (C&A-GTS-QOL) | Assessments will be conducted at baseline, during the treatment phase (weeks 4, 8, and 12), and during the follow-up phase (week 24)
  This scale is specifically designed for patients with Chronic Tic Disorders (CTD) and, compared to generic quality of life instruments, provides a more precise assessment of CTD-related quality of life. The scale comprises 27 items across four domains: Psychological well-being (11 items), Activities of daily living (7 items), Obsessive-compulsive thoughts and behaviors (5 items), Cognitive functioning (4 items).
  Each item is rated using a 5-point Likert scale. Positively worded items are scored from 1 ("strongly disagree") to 5 ("strongly agree"), while reverse-scored items are inversely coded. Domain scores are calculated by summing the item scores within each domain, and the total raw score is derived by aggregating all domain scores.
Child Behavior Checklist (CBCL) | Assessments will be conducted at baseline, during the treatment phase (weeks 4, 8, and 12), and during the follow-up phase (week 24)
  The CBCL evaluates general information, social competence, and behavioral problems.
  Social Competence:
  Encompasses three domains: activities, social interactions, and academic performance.
  Behavioral Problems:
  Assesses 113 items across domains such as depression, anxiety, and aggression.
  Items are scored on a 3-point Likert scale:
  0: Absent
  1. Mild or occasional
  2. Marked or frequent This framework enables a comprehensive evaluation of acupuncture's impact on behavioral outcomes in children with tic disorders by integrating multidimensional metrics of social adaptation and psychopathology.

CONTACTS AND LOCATIONS:
Overall Officials: Hao Zhou, M.D., Principal Investigator — Children's Hospital of Fudan University
Locations (1):
- Children's Hospital, Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
The trial results will be published in a peer-reviewed scientific paper and through oral presentations at conferences. The datasets （IPD） during the current study are available from the corresponding author on reasonable request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be made available for sharing for one year following the publication of the research results as a peer-reviewed paper.
Access Criteria: Data will be available for non-commercial research upon reasonable request to the corresponding author, subject to a signed data use agreement and ethical compliance. Sharing is limited to 1 year post-publication.

REFERENCES:
- [Background] Leckman JF. Tic disorders. BMJ. 2012 Jan 5;344:d7659. doi: 10.1136/bmj.d7659. No abstract available. PMID 22223834
- [Background] Oluwabusi OO, Parke S, Ambrosini PJ. Tourette syndrome associated with attention deficit hyperactivity disorder: The impact of tics and psychopharmacological treatment options. World J Clin Pediatr. 2016 Feb 8;5(1):128-35. doi: 10.5409/wjcp.v5.i1.128. eCollection 2016 Feb 8. PMID 26862512
- [Background] Knight T, Steeves T, Day L, Lowerison M, Jette N, Pringsheim T. Prevalence of tic disorders: a systematic review and meta-analysis. Pediatr Neurol. 2012 Aug;47(2):77-90. doi: 10.1016/j.pediatrneurol.2012.05.002. PMID 22759682
- [Background] Jiang Yanlin, Zhang Qiang, Zhai Rui, Peng Yaqi, Tai Ran, and Wang Junhong. Systematic Review on the Prevalence and Risk Factors of Tic Disorders in Chinese Children. Chinese Journal of Child Health Care. 2023; 31: 661-667.
- [Background] Yang C, Zhang L, Zhu P, Zhu C, Guo Q. The prevalence of tic disorders for children in China: A systematic review and meta-analysis. Medicine (Baltimore). 2016 Jul;95(30):e4354. doi: 10.1097/MD.0000000000004354. PMID 27472724
- [Background] Liu ZS, Cui YH, Sun D, Lu Q, Jiang YW, Jiang L, Wang JQ, Luo R, Fang F, Zhou SZ, Wang Y, Cai FC, Lin Q, Xiong L, Zheng Y, Qin J. Current Status, Diagnosis, and Treatment Recommendation for Tic Disorders in China. Front Psychiatry. 2020 Aug 13;11:774. doi: 10.3389/fpsyt.2020.00774. eCollection 2020. PMID 32903695
- [Background] Yang C, Cheng X, Zhang Q, Yu D, Li J, Zhang L. Interventions for tic disorders: An updated overview of systematic reviews and meta analyses. Psychiatry Res. 2020 May;287:112905. doi: 10.1016/j.psychres.2020.112905. Epub 2020 Mar 1. PMID 32163785
- [Background] Pringsheim T, Okun MS, Muller-Vahl K, Martino D, Jankovic J, Cavanna AE, Woods DW, Robinson M, Jarvie E, Roessner V, Oskoui M, Holler-Managan Y, Piacentini J. Practice guideline recommendations summary: Treatment of tics in people with Tourette syndrome and chronic tic disorders. Neurology. 2019 May 7;92(19):896-906. doi: 10.1212/WNL.0000000000007466. PMID 31061208
- [Background] Kim DD, Barr AM, Chung Y, Yuen JWY, Etminan M, Carleton BC, White RF, Honer WG, Procyshyn RM. Antipsychotic-Associated Symptoms of Tourette Syndrome: A Systematic Review. CNS Drugs. 2018 Oct;32(10):917-938. doi: 10.1007/s40263-018-0559-8. PMID 30121819
- [Background] Roessner V, Eichele H, Stern JS, Skov L, Rizzo R, Debes NM, Nagy P, Cavanna AE, Termine C, Ganos C, Munchau A, Szejko N, Cath D, Muller-Vahl KR, Verdellen C, Hartmann A, Rothenberger A, Hoekstra PJ, Plessen KJ. European clinical guidelines for Tourette syndrome and other tic disorders-version 2.0. Part III: pharmacological treatment. Eur Child Adolesc Psychiatry. 2022 Mar;31(3):425-441. doi: 10.1007/s00787-021-01899-z. Epub 2021 Nov 10. PMID 34757514